CLINICAL TRIAL: NCT02607137
Title: Evaluation of Training Program on Promoting Family Holistic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); Social Welfare Department, Hong Kong (Other Government); Christian Family Service Centre (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Research Officer, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UW 14-601
Record Dates: First submitted 2015-11-14; First posted 2015-11-17 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Health Education (Experimental): Health information related to physical activity
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Health Education — Information on healthy living style in relation to physical activity

SUMMARY:
Holistic health is an integration and interaction of physical and psychosocial health. Positive psychology is a science of happiness, which focuses on positive emotions and personal strengths. It also is crucial component in family holistic health. Healthy diet can help to achieve energy balance and healthy weights. Physical activity is believed to contribute to physical and mental health, as well as social well-being. However, physical inactivity was found to be a local and worldwide issue and most Hong Kong people are having a sedentary lifestyle.

In view of the health challenges locally and globally, the new phase of FAMILY project will focus to promote family holistic health with emphasize on the interaction and integration of physical and psychosocial health. The investigator will initiate and develop a series innovative training program with vigorous evaluation in order to evaluate the effectiveness of the programs. The investigator hypothesize that the training programs would promote the health awareness and the health of the participants

DETAILED DESCRIPTION:
Holistic health is an integration and interaction of physical and psychosocial health. Positive psychology is a science of happiness, which focuses on positive emotions and personal strengths. It is used as a preventive and complementary medicine, which also is crucial component in family holistic health (happiness, harmony and health). Healthy diet can help to achieve energy balance and healthy weights. Sufficient daily consumption of fruit and vegetables, as well as limitation on the intake of sugar, salt and fat could prevent major diseases, such as cardiovascular diseases and certain cancers. Physical activity is believed to contribute to physical and mental health, as well as social well-being. However, physical inactivity was found to be a local and worldwide issue and most Hong Kong people are having a sedentary lifestyle. Studies show that the increase of physical activity and healthy diet reduce the risk of chronic diseases, and improve cardio-pulmonary functions; whereas sedentary behaviors increase the risk

Although people understand the harmful effect of family disharmony, physical inactivity and unhealthy diet, which may cause different kinds of physical and mental illnesses, healthy living attitudes and behaviours are lacking.

Over the past six years, the FAMILY project has been working on community-based projects to promote FAMILY health, happiness and harmony (3Hs). In view of the health challenges locally and globally, the new phase of FAMILY project will put more emphasis on health in the upcoming three years. Following the theme on FAMILY 3Hs, the new work focus is to promote family holistic health with emphasize on the interaction and integration of physical and psychosocial health. The investigator will initiate and develop a series innovative community-based projects and training program with vigorous evaluation in order to evaluate the effectiveness of the programs.

The investigator hypothesize that the training programs would promote the health awareness and the health of the participants. During the training, the investigator will conduct physical fitness test and collect data from the participants. Those participants would conduct community programmes for their own institution to enhance the personal and family well-being of their service users.

In order to assess the effectiveness of the training program on improving individual and family well-being and their capability of community programme implementation, Self-reported questionnaire would be used at baseline, one month and three months after training; and focus group interview would be conducted after participants finishing their community programmes.

ELIGIBILITY:
Inclusion Criteria:

* Chinese speaking
* able to complete study questionnaire
* aged 18 or above

Exclusion Criteria:

* not fit the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in health behavior in relation to physical activity | Baseline , 1 month
  Change in health behavior in relation to physical activity will be assessed by behavior indicator scale

SECONDARY OUTCOMES:
Changes in knowledge and attitude on performing physical activity | Baseline, 1 month and 3 months
  Change in knowledge and attitude on performing physical activity will be assessed by outcome-based questionnaire
Change in subjective happiness | Baseline, 1 month and 3 months
  Subjective happiness will be assessed by outcome-based questionnaire
Change in family health, happiness and harmony (Family 3Hs) | Baseline, 1 month
  Family 3Hs will be assessed by family well-being scale
Change in Quality of Life | Baseline, 1 month and 3 months
  Change in quality of life will be assessed by SF-12 v2 health survey
Changes in physical fitness | Baseline, 1 month and 3 months
  Change in physical fitness will be assessed by simple fitness test
Changes in health behavior in relation to physical activity | Baseline, 1 month and 3 months
  Change in health behaviour will be assessed by behavior indicator scale
Change in family communication in relation to Zero Time Exercise | Baseline, 1 month, 3 months
  Change in family communication will be assessed by behavior indicator scale
Reactions to training content | Immediately after finishing training workshop "up to 30 min"
  Assessed by outcome-based questionnaire
Learning in relation to implementing community programmes | Baseline, 1 month, 3 months
  Assessed by outcome-based questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Lai, DN, Principal Investigator — The University of Hong Kong
Locations (1):
- The Boys' & Girls' Association of Hong Kong, Wan Chai, Hong Kong

REFERENCES:
- [Background] Bellicha A, Kieusseian A, Fontvieille AM, Tataranni A, Charreire H, Oppert JM. Stair-use interventions in worksites and public settings - a systematic review of effectiveness and external validity. Prev Med. 2015 Jan;70:3-13. doi: 10.1016/j.ypmed.2014.11.001. Epub 2014 Nov 10. PMID 25449692
- [Background] Gardiner PA, Eakin EG, Healy GN, Owen N. Feasibility of reducing older adults' sedentary time. Am J Prev Med. 2011 Aug;41(2):174-7. doi: 10.1016/j.amepre.2011.03.020. PMID 21767725
- [Background] Torbeyns T, Bailey S, Bos I, Meeusen R. Active workstations to fight sedentary behaviour. Sports Med. 2014 Sep;44(9):1261-73. doi: 10.1007/s40279-014-0202-x. PMID 24842828
- See also: Fact Sheet on Physical Activity — http://www.who.int/mediacentre/factsheets/fs385/en/
- See also: GovHK: Exercise and Nutrition — http://www.gov.hk/en/residents/health/healthadvice/healthcare/exercise.htm